CLINICAL TRIAL: NCT06884371
Title: Is a Complete Fatty Infilteration of Lumbar Paraspinal Muscles an Indicator to a Serious Pathology: A Case Report
Brief Title: Lumbar Paraspinal Muscle Fatty Infilteration
Status: Completed | Type: Observational
Sponsor: Noha Khaled Shoukry (Other)
Responsible Party: Sponsor-Investigator, Noha Khaled Shoukry, doctor, Cairo University
Organization: Cairo University (Other)
Other Study IDs: cairo university PT 1
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Muscle Weakness
MeSH Terms: conditions — Muscle Weakness | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: physical therapy — ultrasound and TENS for the back

SUMMARY:
Introducing a unique clinical case of limb-girdle muscular dystrophy associated with LBP that was initially misdiagnosed as non-specific LBP

DETAILED DESCRIPTION:
This case report describes the history, examination findings, and clinical reasoning used for a patient suffering from LBP as a chief complaint. A new sign appeared in MRI, which prompted the author to change the diagnosis process from lower back pain to a mysterious neurological disease, The MRI revealed widespread fat deposit in the lumbar paraspinal muscles. This MRI sign prompted the authors to do more lab investigation, showing a notably elevated level of creatinine phosphokinase (906 u/L). Further clinical examination revealed proximal muscle weakness, winging of scapula and Bilateral LMN facial palsy. Therefore, the patient was ultimately directed to a neurologist who confirmed the diagnosis of limb-girdle muscular dystrophy

ELIGIBILITY:
Inclusion Criteria:

* experiencing lower back stiffness and a dull back pain

Exclusion Criteria:

* diabetes, heart disease, or muscle disease. any history of previous falls, accidents, surgeries, hospitalizations, and he denied any significant past illnesses, or allergies.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: A 22-year-old man who used to work eight hours a day sitting for a long time in an office
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
An MRI of the lumbar spine | one month

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided